CLINICAL TRIAL: NCT02700438
Title: Perianal Application of Glyceryl Trinitrate 0.4% Ointment vs Percutaneous Posterior Tibial Nerve Stimulation in the Treatment of Chronic Anal Fissure
Brief Title: Glyceryl Trinitrate Ointment vs Posterior Tibial Nerve Stimulation in the Treatment of Anal Fissure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, MD, PhD, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CG15-02
Record Dates: First submitted 2016-02-25; First posted 2016-03-07 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glyceryl trinitrate ointment (Active Comparator): Commercially available aluminium tubes containing 0.4 glyceryl trinitrate ointment (Rectogesic, proStrakan Group, Galashiels, UK) were purchased from pharmacies. The dosage for all the patients was 375 mg of ointment (containing 1.5 mg of glyceryl trinitrate), applied with a gloved finger to the distal anal canal, every 12 hours for an 8-week period.
  Interventions: Drug: Glyceryl trinitrate ointment
- Urgent PC Neuromodulation System® (Experimental): The Urgent PC Neuromodulation System® (Uroplasty, Minnetonka, MN, USA) was used for percutaneous posterior tibial nerve stimulation. Subjects underwent one 30-min session 2 days per week for 8 consecutive weeks in an outpatient clinic. Patients were placed in the supine position without anesthesia. PPTNS was delivered using a needle electrode that was inserted 3-4cm cephalad and 2 cm posterior to the medial malleolus at a 60º angle towards the ankle joint to a depth of approximately 0.5-1cm. Successful placement was confirmed by the presence of electric sensation 5 cm above and below the insertion site or a digital plantar flexion. PPTNS was undertaken at the highest amplification (0-20 mA) at a frequency of 20 Hz, causing neither a motor response nor pain.
  Interventions: Procedure: Urgent PC Neuromodulation System®

INTERVENTIONS:
Drug: Glyceryl trinitrate ointment — Application of 375 mg of ointment to the distal anal canal, every 12 hours for an 8-week period.
  Other Names: Rectogesic
  Arms: Glyceryl trinitrate ointment
Procedure: Urgent PC Neuromodulation System® — Subjects underwent one 30-min session of percutaneous posterior tibial nerve stimulation 2 days per week for 8 consecutive weeks in an outpatient clinic, with a Urgent PC Neuromodulation System®. Patients were placed in the supine position without anesthesia. PPTNS was delivered using a needle electrode that was inserted 3-4cm cephalad and 2 cm posterior to the medial malleolus at a 60º angle towards the ankle joint to a depth of approximately 0.5-1cm. Successful placement was confirmed by the presence of electric sensation 5 cm above and below the insertion site or a digital plantar flexion.
  Other Names: PTNS
  Arms: Urgent PC Neuromodulation System®

SUMMARY:
A prospective randomized study was performed. Compliance with the treatment and healing rate of chronic anal fissure in patients receiving glyceryl trinitrate ointment (GTO) and subjects undergoing percutaneous posterior tibial nerve stimulation (PPTNS) were evaluated .

DETAILED DESCRIPTION:
Patients were randomly assigned to experimental and control groups: those patients undergoing PPTNS (Experimental Group - EG) and those receiving glyceryl trinitrate ointment (Control Group - CG).

Treatments:

Glyceryl trinitrate ointment (GTO): Commercially available aluminium tubes containing 0.4 glyceryl trinitrate ointment (Rectogesic, proStrakan Group, Galashiels, UK) were purchased from pharmacies. The dosage for all the patients was 375 mg of ointment (containing 1.5 mg of glyceryl trinitrate), applied with a gloved finger to the distal anal canal, every 12 hours for an 8-week period.

PPTNS: The Urgent PC Neuromodulation System® (Uroplasty, Minnetonka, MN, USA) was used. Subjects underwent one 30-min session 2 days per week for 8 consecutive weeks in an outpatient clinic. Patients were placed in the supine position without anesthesia. PPTNS was delivered using a needle electrode that was inserted 3-4cm cephalad and 2 cm posterior to the medial malleolus at a 60º angle towards the ankle joint to a depth of approximately 0.5-1cm. Successful placement was confirmed by the presence of electric sensation 5 cm above and below the insertion site or a digital plantar flexion. PPTNS was undertaken at the highest amplification (0-20 mA) at a frequency of 20 Hz, causing neither a motor response nor pain.

Compliance with the treatment and healing rate of chronic anal fissure was investigated.

ELIGIBILITY:
Inclusion Criteria:

* persistent anal fissure after the failure of hygienic and dietary measures over at least a 6-week period

Exclusion Criteria:

* associated anal pathologies
* intestinal inflammation disorders
* fissures secondary to underlying diseases
* patients with previous history of headaches

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of participants who discontinued the assigned treatment | 8 weeks
  The discontinuity with each treatment will be evaluated by means of face-to-face interviews in the Outpatient Clinic every week, investigating the compliance with the prescribed therapy (correct administration of the ointment and performance of the percutaneous posterior tibial nerve stimulation sessions). The number of patients who stop the therapy will be considered as a treatment withdrawal.

SECONDARY OUTCOMES:
Healing, defined as disappearance of symptoms and evidence of fissure reepithelization | 8 weeks
  Healing will be defined as disappearance of symptoms and evidence of fissure reepithelization

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Barna, MD, PhD, Study Chair — Garcilaso Clinic

IPD SHARING:
Plan to Share IPD: Yes